CLINICAL TRIAL: NCT05980065
Title: A Dose-block Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose, First-in-human, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics After Subcutaneous Administration of C1K in Healthy Subjects
Brief Title: To Evaluate the Safety, Tolerability, and Pharmacokinetics After Subcutaneous Administration of C1K in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ensol Biosciences, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C1K-101
Record Dates: First submitted 2023-04-19; First posted 2023-08-07 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2022-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose level 1 (Experimental): C1K 150mg
  Interventions: Drug: C1K
- Dose level 2 (Experimental): C1K 300mg or placebo
  Interventions: Drug: C1K; Drug: Placebo
- Dose level 3 (Experimental): C1K 600mg or placebo
  Interventions: Drug: Placebo; Drug: C1K
- Dose level 4 (Experimental): C1K 900mg or placebo
  Interventions: Drug: Placebo; Drug: C1K
- Dose level 5 (Experimental): C1K 1200mg or placebo
  Interventions: Drug: Placebo; Drug: C1K

INTERVENTIONS:
Drug: C1K — Subcutaneously administrate C1K 150mg at 0 Day 1, Day 8, Day 15
  Arms: Dose level 1
Drug: C1K — Subcutaneously administrate C1K 300mg at 0 Day 1, Day 8, Day 15
  Arms: Dose level 2
Drug: Placebo — Subcutaneously administrate placebo at 0 Day 1, Day 8, Day 15
  Arms: Dose level 2; Dose level 3; Dose level 4; Dose level 5
Drug: C1K — Subcutaneously administrate C1K 600mg at 0 Day 1, Day 8, Day 15
  Arms: Dose level 3
Drug: C1K — Subcutaneously administrate C1K 900mg at 0 Day 1, Day 8, Day 15
  Arms: Dose level 4
Drug: C1K — Subcutaneously administrate C1K 1200mg at 0 Day 1, Day 8, Day 15
  Arms: Dose level 5

SUMMARY:
A dose-block randomized, double-blind, placebo-controlled, single and multiple ascending dose, first-in-human, phase 1 first in human clinical trial to evaluate the safety, tolerability, and pharmacokinetics after subcutaneous administration of C1K in healthy Korean subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 19 - 45 years at the time of screening visit procedure.
2. The subject weighs in the range of 50.0 - 90.0 kg and has a body mass index (BMI) in the range 18-27 kg/m2.
3. Sufficient ability to understand the study after being informed about the study and provide written informed consent.
4. Based on physical examination, vital sign, 12-lead ECG and laboratory test etc. and in the opinion of the investigator, the subject is suitable for the study.

Exclusion Criteria:

1. A subject with clinically significant hepatobiliary, renal, neurologic, respiratory, endocrine, blood•oncology, cardiovascular, urinary, or, psychical diseases or a history
2. A subject who has difficulty with sub-cutaneous injection(ex: tattoo, allergy on skin etc.)
3. A subject who has hypersensitivity to the drugs of the drugs containing the same class, or other drugs, or a history of clinically significant hypersensitivity
4. A subject who has ventricular tachycardia, ventricular tachycardia, ventricular flutter or confirmed other ventricular flutter and QTc interval: > 450 ms or the other clinically significant medical findings
5. A subject with the following results in the screening test:

   * Blood AST (GOT), ALT (GPT): > Normal range upper × 1.5
   * Blood CPK > Normal range upper × 1.5
   * eGFR (CKD-EPI equation) < 60 mL/min/1.73 m2
6. Positive serological test (syphilis test, hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test)
7. A subject with the following results in the screening test:

   * systolic blood pressure < 80 mmHg or > 140 mmHg
   * diastolic blood pressure < 50 mmHg or > 90 mmHg
8. A subject with a history of drug abuse or positive urine screening test for drug abuse
9. A subject who administered any prescription drugs or herbal medicine within 2 weeks prior to the expected date of the first dose, or any over-the-counter drug (OTC drug) or vitamin within 1 week prior to the expected date of the first dose (However, can participate in the study if otherwise decided eligible by the investigator).
10. A subject who participated in other clinical trial and administered investigational drug within 6 months prior to the expected date of the first dose
11. A subject who donated whole blood within 2 months or the component blood within 1 month prior to the expected date of the first dose, or received blood transfusion within 1 month prior to the expected date of the first dose
12. Smokers who smoke more than 10 cigarettes/day in the last 3 months as of screening day.
13. A subject with persistent alcohol intake (> 21 units/week, 1 unit = 10 g of pure alcohol), or inability to abstain from drinking from 3 days before the expected date of the first dose until the last discharge
14. A male subject who has plan to have a baby or to donate sperm. A female subject who is pregnant or lactating or has plan to lactate within 3 months after administration of IP
15. A subject who is intending to become pregnant during this study or with inability to use a medically acceptable contraception method(ex. sterilization operation, intrauterine device etc. for Subject or subject's partner

    ※ medically acceptable contraception method
    * Use of intrauterine device which is proven pregnancy failure rates in spouses (or partners).
    * Use combined blocking contraceptives (for male or female) and antiseptic drugs
    * Subject or partner's operation(vasectomized, bilateral tubal occlusion, hysterectomy)
16. Subject who is considered inadequate to participation in the study due to other reason under investigator's discretion

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Safety assessment by adverse event monitoring | up to 23 days
  Monitoring of adverse event
Cmax | At day 1
  Peak Plasma Concentration
Cmax | At day 15
  Peak Plasma Concentration
AUC | At day 1
  Area under the plasma concentration versus time curve
AUC | At day 15
  Area under the plasma concentration versus time curve

SECONDARY OUTCOMES:
Safety-Injection site response evaluation | up to 23 days
  To evaluate safety
Systolic blood pressure | up to 23 days
  Monitoring of vital signs
Diastolic blood pressure | up to 23 days
  Monitoring of vital signs
Pulse rate | up to 23 days
  Monitoring of vital signs
QT interval | up to 23 days
  Monitoring of 12-lead electrocardiogram
QTc interval | up to 23 days
  Monitoring of 12-lead electrocardiogram
PR interval | up to 23 days
  Monitoring of 12-lead electrocardiogram
QRS interval | up to 23 days
  Monitoring of 12-lead electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: JAESEONG OH, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No